CLINICAL TRIAL: NCT03893123
Title: Prostate Cancer Risk in Firefighters: Its Association to Qualitative and Quantitative Indicators of Exposure
Brief Title: Prostate Cancer Risk in Firefighters
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Institute of Public Health (Other Government); Extrastiftelsen (Other); National Institute of Occupational Health (Unknown); Norwegian Confederation of Trade Unions (Unknown); Fagforbundet (Unknown); Gjensidige Foundation (Unknown); Norwegian Cancer Society (Other); Norwegian Firefighters Fight Cancer (Unknown); Norwegian Labour Inspection Authority (Unknown)
Responsible Party: Principal Investigator, Jarle Jakobsen, PhD-student, Norwegian Institute of Public Health
Other Study IDs: 2016/2282
Record Dates: First submitted 2019-03-25; First posted 2019-03-28 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Prostatic Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Firefighters
  Interventions: Other: Observational study, prostate cancer is outcome of interest

INTERVENTIONS:
Other: Observational study, prostate cancer is outcome of interest — Observational study

SUMMARY:
Firefighters have been shown to be at increased risk for various types of cancer, including prostate cancer. This study will try to explore possible reasons for this increase in risk. A study group at the Cancer Registry of Norway is creating a cohort of Norwegian firemen employed from 1960 onwards. A job exposure matrix (JEM) is also being constructed, examining different types of exposure to potentially cancer-inducing agents and activities, and how these have changed historically. Examples include exposure to fire-smoke, shiftwork, diesel exhaust and regular health check-ups. By linking the cohort with data from the Cancer Registry of Norway and the JEM the investigators can examine which exposure assessments, if any, are related to an increased risk of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Work as firefighter as recorded by the participating fire stations

Exclusion Criteria:

* Any other occupation, including chimney sweepers

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Norwegian males
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of prostate cancer | From January 1st 1960 until December 31st 2018
  As reported to the Cancer Registry of Norway

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Registry of Norway, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No